CLINICAL TRIAL: NCT04770519
Title: Genetic Studies of Strabismus, Nystagmus, and Associated Disorders
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Mary Whitman, Associate Professor of Ophthalmology, Boston Children's Hospital
Other Study IDs: IRB-P00036313; R01EY032539 (NIH)
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Strabismus; Nystagmus, Congenital
Keywords: strabismus; esotropia; exotropia; nystagmus
MeSH Terms: conditions — Strabismus; Nystagmus, Congenital; Esotropia; Exotropia; Nystagmus, Pathologic | interventions — Whole Genome Sequencing; Exome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: whole genome sequencing or whole exome sequencing — Whole genome sequencing or whole exome sequencing will be performed for all enrolled participants.

SUMMARY:
Strabismus (misalignment of the eyes) often runs in families. In this study, the investigators are looking for genetic variants associated with strabismus and nystagmus. Three types of subects will be enrolled: (1) Families with at least 3 members with strabismus, (2) individuals with infantile esotropia and their parents and siblings, and (3) individuals with infantile nystagmus and their parents. Whole exome and/or whole genome sequencing will be used to identify genetic variants shared by family members with strabismus and to identify genetic causes of nystagmus.

ELIGIBILITY:
Inclusion Criteria:

- Member of a family with at least 3 biological relatives with strabismus. (Both affected and non-affected family members will be enrolled).

OR

- Member of a family with at least 1 individual with infantile esotropia. (Both affected and non-affected family members will be enrolled).

OR

- Member of a family with at least 1 individual with infantile nystagmus. (Both affected and non-affected family members will be enrolled).

Exclusion Criteria:

* paralytic strabismus in affected family members

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All willing members of families in which 3 or more biological relatives have strabismus (esotropia, exotropia, or vertical misalignments) with full eye movements, or affected individual has infantile esotropia or infantile nystagmus.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants | 2 years
  genetic variants shared by family members with strabismus

CONTACTS AND LOCATIONS:
Overall Officials: Mary Whitman, MD/PhD, Principal Investigator — Assistant Professor
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified genetic data will be deposited in dbGAP (database of genotypes and phenotypes) after publication.
Time Frame: At time of publication
Access Criteria: de-identified data will be available per dbGAP access policies.